CLINICAL TRIAL: NCT04105374
Title: A Phase II/III Randomized, Open-Label Study of Toca 511, A Retroviral Replicating Vector, Combined With Toca FC With Temozolomide and Radiation Followed by Adjuvant Temozolomide and Toca FC Compared to Temozolomide and Radiation Followed by Adjuvant Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Testing the Addition of an Anti-cancer Viral Gene Therapy, Toca 511/Toca FC, to the Usual Treatment (Temozolomide and Radiation Therapy) for Newly Diagnosed Glioblastoma
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: NCI approval withdrawn
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BN006; NCI-2019-04562 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN006 (Other: NRG Oncology); NRG-BN006 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Anaplastic Astrocytoma; Glioblastoma; Oligodendroglioma; Supratentorial Glioblastoma
Keywords: Toca 511; Toca FC
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Oligodendroglioma | interventions — Radiotherapy; Radiation; Temozolomide; vocimagene amiretrorepvec; DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (surgery, radiation therapy, temozolomide) (Active Comparator): Beginning on week 5 following standard of care surgery, patients undergo radiation therapy over 30 fractions 5 days per week for up to 6 weeks, and receive temozolomide PO QD for up to 49 days. At the discretion of treating physician, patients may also receive novoTTF-100A (Optune) device 0-7 weeks following radiation and temozolomide treatment. One month following completion of radiation therapy, patients continue to receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: NovoTTF-100A Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Temozolomide; Procedure: Therapeutic Conventional Surgery
- Arm II (Toca 511, Toca FC, radiation therapy, temozolomide) (Experimental): Patients receive vocimagene amiretrorepvec via intracranial injection during surgery on day 1. Beginning on week 5 following surgery, patients receive extended release flucytosine PO TID for 7 consecutive days every 7 weeks. Patients also undergo radiation therapy and receive temozolomide as in arm I. After completion of radiation therapy and at the discretion of the treating physician, patients may continue to receive extended release flucytosine PO TID for 7 consecutive days every 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Extended Release Flucytosine; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Temozolomide; Procedure: Therapeutic Conventional Surgery; Biological: Vocimagene Amiretrorepvec

INTERVENTIONS:
Drug: Extended Release Flucytosine — Given PO
  Other Names: Extended Release 5-FC; Extended Release 5-Fluorocytosine; Extended-Release 5-FC; Extended-Release 5-Fluorocytosine; Extended-Release Flucytosine; Toca FC
  Arms: Arm II (Toca 511, Toca FC, radiation therapy, temozolomide)
Device: NovoTTF-100A Device — Receive Optune device
  Other Names: NovoTTF-100A; NovoTTF-100A System; NovoTTFields; NovoTumor Treatment Fields; Optune; Optune Device
  Arms: Arm I (surgery, radiation therapy, temozolomide)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery
Biological: Vocimagene Amiretrorepvec — Given via intracranial injection
  Other Names: DNA (Synthetic Toca 511-encoding Retroviral Vector AC3-yCD2(V)); Toca 511
  Arms: Arm II (Toca 511, Toca FC, radiation therapy, temozolomide)

SUMMARY:
This phase II/III trial studies how well vocimagene amiretrorepvec (Toca 511) and extended release flucytosine (Toca FC) work when added to the usual treatment (temozolomide and radiation therapy) in treating patients with newly diagnosed glioblastoma. Toca 511 is a live virus that has been built to carry a gene into tumor cells. This gene carries instructions that cause the tumor cells to turn Toca FC, typically used to treat fungal infections, into a drug that may kill the tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving Toca 511 and Toca FC in addition to the usual treatment (temozolomide and radiation therapy) may help shrink or stabilize cancer or extend the life of patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival (PFS) of patients with newly diagnosed glioblastoma treated with Toca 511 at the time of tumor resection followed by Toca FC in combination with standard of care (SOC) treatment to patients with newly diagnosed glioblastoma treated with SOC after tumor resection. (Phase II) II. To compare the overall survival (OS) from time of randomization of all patients with newly diagnosed glioblastoma treated with Toca 511 at the time of tumor resection followed by Toca FC in combination with SOC treatment to patients with newly diagnosed glioblastoma treated with SOC after tumor resection. (Phase III)

SECONDARY OBJECTIVES:

I. To evaluate the safety of each arm as administered in this study. II. To compare the OS between arms (only for phase II part of the study). III. To compare the PFS between arms using Response Assessment in Neuro-Oncology (RANO) (only for phase III part of the study).

IV. To evaluate the objective response rate (ORR) in patients with measurable disease at the post-surgical scan.

V. To evaluate the effect of IDH mutation status on survival outcomes between arms.

VI. To evaluate the PFS and OS by extent of resection. VII. To evaluate the effect of MGMT methylation status on survival outcomes between arms.

EXPLORATORY OBJECTIVES:

I. To evaluate the duration of response (DoR) in patients with measurable disease at the post-surgical scan using mRANO.

II. To evaluate the effect of corticosteroids administration on efficacy of Toca 511 and Toca FC.

III. To optimize quality assurance methodologies and processes for radiotherapy and imaging.

IV. To determine if there is a tumor-microenvironment signature based on ribonucleic acid (RNA) sequencing that is associated with a selective increase in benefit from the addition of Toca 511 and Toca FC.

V. To compare regional genomic heterogeneity and molecular profiles, as measured by RNA sequencing and methylation analyses between arms.

VI. To compare quality of life (QOL), as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) and Brain Cancer Module (BN20), between arms.

VII. To compare health utilities, as measured by the EuroQoL 5-Dimension 5-Level (EQ-5D-5L), between arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Beginning on week 5 following standard of care surgery, patients undergo radiation therapy over 30 fractions 5 days per week for up to 6 weeks, and receive temozolomide orally (PO) once daily (QD) for up to 49 days. At the discretion of treating physician, patients may also receive novoTTF-100A (Optune) device 0-7 weeks following radiation and temozolomide treatment. One month following completion of radiation therapy, patients continue to receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive vocimagene amiretrorepvec via intracranial injection during surgery on day 1. Beginning on week 5 following surgery, patients receive extended release flucytosine PO three times daily (TID) for 7 consecutive days every 7 weeks. Patients also undergo radiation therapy and receive temozolomide as in arm I. After completion of radiation therapy and at the discretion of the treating physician, patients may continue to receive extended release flucytosine PO TID for 7 consecutive days every 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up until progression then, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Presumptive diagnosis of glioblastoma based on magnetic resonance imaging (MRI) imaging within 14 days prior to registration.

  * NOTE: Patients who undergo treatment with Toca 511 whose final pathology shows diagnosis other than glioblastoma (e.g. anaplastic astrocytoma or oligodendroglioma or any other histology) will be treated with Toca FC and chemoradiation; however they will not be analyzed in the primary endpoint. The outcomes of these patients will be reported descriptively. Similarly the patients with anaplastic astrocytoma or oligodendroglioma or any other histology treated on the standard-of-care arm will be reported separately and they are allowed to receive the treatment per choice of the treating physician/ investigator (for e.g. radiation therapy [RT] plus temozolomide or RT plus procarbazine-lomustine-vincristine [PCV])
* In addition, patients who have undergone biopsy with diagnosis of glioblastoma and who have never received any chemotherapy and/or radiation and are candidates for >= 80% resection of enhancing region are eligible
* The tumor must be unifocal, confined to the supratentorial compartment and based on the pre-operative evaluation, the patient is a candidate for >= 80% resection of enhancing region
* Measurable disease preoperatively, defined as at least 1 contrast enhancing lesion, with 2 perpendicular measurements of at least 1 cm, as per Response Assessment in Neuro-Oncology (RANO) criteria
* The hematoxylin and eosin (H&E) slide and formalin-fixed paraffin-embedded (FFPE) tumor tissue block must be available to be sent for mandatory central pathology review after registration
* Patients must be able to undergo an evaluation by MRI within 96 hours post surgery to assess extent of resection
* Karnofsky performance status >= 70 within 14 days prior to registration
* History/physical examination within 14 days prior to registration
* Platelet count >= 100,000/mm^3 (within 14 days prior to registration)
* Hemoglobin (Hgb) >= 10 g/dL (within 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (within 14 days prior to registration)
* Absolute lymphocyte count (ALC) >= 1000/mm^3 (within 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless has Gilbert?s syndrome) (within 14 days prior to registration)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (within 14 days prior to registration)
* Estimated glomerular filtration rate of at least 50 mL/min by the Cockcroft Gault formula (within 14 days prior to registration)
* Women of childbearing potential (women who have not had >=12 months of non therapy induced amenorrhea or are not surgically sterile) must have had a negative serum pregnancy test within 14 days prior to registration and must agree to use a birth control method in addition to barrier methods (condoms or diaphragm) during treatment with temozolomide
* If the patient is randomized to arm 2, the patient or patient?s partner must be willing to use barrier method of contraception for 12 months after receiving Toca 511 and 1 month after stopping Toca FC or until there is no evidence of the virus in the patient?s blood, whichever is longer
* The patient or a legally authorized representative must provide study-specific informed consent prior to registration

Exclusion Criteria:

* History of prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* A contrast enhancing brain tumor on MRI that is any of the following:

  * Multi focal (defined as 2 separate areas of contrast enhancement measuring at least 10 mm in 2 planes that are not contiguous on either fluid attenuated inversion recovery [FLAIR] or T2 hyperintensity);
  * Associated with either diffuse subependymal or leptomeningeal dissemination; or
  * > 50 mm in any dimension
* Active infection (excluding skin or toenail infections) requiring systemic antibiotic, antifungal or antiviral therapy within 28 days prior to registration
* Bleeding diathesis, or must take anticoagulants, or antiplatelet agents, including nonsteroidal anti inflammatory drugs (NSAIDs), at the time of the scheduled resection that cannot be stopped for surgery
* Known human immunodeficiency virus (HIV) positive status
* History of allergy or intolerance to flucytosine
* Swallowing difficulty that would prevent patient from being able to swallow either temozolomide or Toca FC or severe active mal-absorption
* Patients who are breast feeding or lactating
* Intent to undergo treatment with the Gliadel wafer at the time of this surgery or has received the Gliadel
* Prior to registration, steroid treatment beyond a maximum of 8 mg/day of dexamethasone (or equivalent) or a total of 8 weeks (56 days) is excluded
* Severe pulmonary, cardiac or other systemic disease, specifically:

  * New York Heart Association > =Class II congestive heart failure within 6 months (180 days) prior to registration, unless asymptomatic and well controlled with medication
  * Uncontrolled or significant cardiovascular disease, clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes), clinically significant pulmonary disease (such as >= grade 2 dyspnea)
  * Any other disease that as per investigator assessment may affect the patient?s compliance or place the patient at higher risk of potential treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Phase II) | Time from randomization to the first documented progressive disease (PD) as determined by central review, or death due to any cause, whichever occurs first, assessed for up to 5 years
  Analysis of treatment comparison between the experimental and standard-of-care arms will be performed once the required number of centrally-reviewed PFS events is reached . The Kaplan-Meier method will be used to calculate the PFS rates for each of the two arms. Hazard ratio (HR) on the treatment effect will be calculated using the stratified Cox proportional hazard model. A one-sided stratified log-rank test will be used to test the difference in PFS between the two arms.
Overall survival (OS) (Phase III) | The time from randomization to death due to any cause, assessed up to 5 years
  Analysis of the treatment comparison between the experimental and standard of care arms will be performed once the required number of deaths is reached. The Kaplan-Meier method will be used to calculate the OS rates for each of the two arms. The primary endpoint will be assessed using a one-sided stratified log-rank test, incorporating only stratification factors, to test the difference in OS between the two arms. Hazard ratio (HR) on the treatment effect will be calculated using the stratified Cox proportional hazard model adjusting for stratification factors. In addition to assessing the effect of treatment arm, IDH mutation status, MGMT status, the interaction between MGMT status and treatment arm, extent of resection, and use of Optune (in only the standard-of-care arm) will be assessed using a log-rank test and Cox proportional hazards models.

SECONDARY OUTCOMES:
Incidence of grade 3 or higher adverse events | Until death, assessed up to 5 years
  Will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Counts of all adverse events (AEs) by grade will be provided by treatment arm. Frequencies and percentages will be provided for the worst grade AE experienced by the patient by treatment arm. The number of patients with at least 1 grade 3 or higher AE will be compared between the treatment arms. A comparison between treatment arms of grade 3 and higher AEs related to any aspect of protocol treatment will be tested. A comparison between arms of the following events will also be conducted: any new solid tumor, hematologic malignancy or myelodysplastic syndrome and any neurologic decline not attributed to tumor progression, and any toxicity that is possibly, probably or definitely related to protocol treatment. All comparisons will be tested using a chi-square test with a two-sided significance level of 0.05.
Overall survival (OS) (Phase II) | The time from randomization to death due to any cause, assessed up to 5 years
  The Kaplan-Meier method will be used to calculate the OS rates for each arm. HR on the group variable will be calculated using the Cox proportional hazard model. A two-sided stratified log-rank test will be used to test the difference in OS and PFS between the two arms at a significance level of 0.05.
Progression free survival (PFS) (Phase III) | Time from randomization to the first documented PD as determined by central review, or death due to any cause, whichever occurs first, assessed for up to 5 years
  The Kaplan-Meier method will be used to calculate the PFS rates for the following sets of groups: treatment arms, IDH mutation status, or extent of resection. HR on the group variable will be calculated using the Cox proportional hazard model. A two-sided stratified log-rank test will be used to test the difference in OS and PFS between the two arms at a significance level of 0.05. In addition to assessing the effect of treatment arm, IDH mutation status, MGMT status, the interaction between MGMT status and treatment arm, extent of resection, and use of Optune (in only the standard-of-care arm) will be assessed using a log-rank test and Cox proportional hazards models.
Objective response rate (ORR) | Up to 18 months
  Will be determined centrally. Frequencies and percent of responses will be provided for each group (treatment arm and IDH mutation status) for patients with measurable disease. Patients with a confirmed complete response (CR) or partial response (PR) will be considered responders. The percent of responders at 1 year will be of interest, although ORR will be calculated at 6 and 18 months as well. Between arm comparisons will be tested using a two-sided chi-square test with a significance level of 0.05.

OTHER OUTCOMES:
Duration of response (DOR) | The duration in which a durable response is observed, spanning from time of initial response until PD, assessed for up to 5 years
  Will only be performed in the subset of patients with measurable disease at the post-surgical MRI who respond per central review using mRANO . The Kaplan-Meier method will be used to estimate the time from initial response to PD with a log rank test used to compare between arm differences. Between arm comparisons will be tested using a t-test or Wilcoxon test, depending on the normality of the data.
Tumor-microenvironment signature | Up to 5 years
  The microenvironmental and tumor signatures are derived from ribonucleic acid (RNA) sequencing. They are continuous variables and will be correlated with tumor response and treatment effect. Descriptive statistics will be provided by treatment arm.
Genome-wide deoxyribonucleic acid (DNA) methylation and copy number profiles | Up to 5 years
  DNA methylation profiles, with the application of the DKFZ classifier, has proven useful to confirm histopathologic diagnosis, identify clinically relevant tumor subtypes and reveal specific DNA copy number changes (for example EGFR amplification in glioblastoma [GBM]). These represent both continuous and categorical variables and will be correlated with tumor response and treatment effect. Descriptive statistics will be provided by treatment arm.
Corticosteroid administration | Up to 5 years
  Corticosteroid administration will be assessed at baseline and throughout treatment and follow-up. Between arm comparisons will be tested using a two-sided chi-square test. Dexamethasone or equivalent dose will also be compared between treatment arms using a t-test or Wilcoxon test, depending on the normality of the data. Time points of interest are pre-treatment, start of chemo radiation therapy (RT), completion of chemo RT, then annually in conjunction with follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet S Ahluwalia, Principal Investigator — NRG Oncology